CLINICAL TRIAL: NCT04478318
Title: Quantitative Comparison of Imaging Characteristics of uEXPLORER and Conventional PET/CT in Patients With Lung Cancer, Lymphoma, and Melanoma Undergoing Standard-of-Care FDG-PET/CT for Initial Staging
Brief Title: Comparison of Imaging Characteristics of uEXPLORER and Conventional PET/CT in Patients With Lung Cancer, Lymphoma, and Melanoma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1506448; CCRD039 (Other: UC Davis Cancer Center)
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Lung Neoplasm; Lymphoma; Melanoma; Fluorodeoxyglucose; Positron-emission Tomography
MeSH Terms: conditions — Lung Neoplasms; Lymphoma; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- uEXPLORER/mCT (Experimental): Each patient will undergo a scan on a total-body PET/CT scanner (uEXPLORER) and then undergo an additional scan on a conventional PET/CT scanner (mCT). The first scan will take place 60 minutes after injection with 18F-FDG and the second scan will be 90 minutes after injection with 18F-FDG.
  Interventions: Device: uEXPLORER/mCT
- mCT/uEXPLORER (Experimental): Each patient will undergo a scan on a conventional PET/CT scanner (mCT) and then undergo an additional scan on a total-body PET/CT scanner (uEXPLORER) . The first scan will take place 60 minutes after injection with 18F-FDG and the second scan will be 90 minutes after injection with 18F-FDG.
  Interventions: Device: mCT/uEXPLORER

INTERVENTIONS:
Device: uEXPLORER/mCT — Participants will undergo a total-body PET/CT scan with the uEXPLORER scanner first, followed by a PET/CT scan with the conventional mCT PET/CT scanner.
  Arms: uEXPLORER/mCT
Device: mCT/uEXPLORER — Participants will undergo a PET/CT scan with the conventional mCT PET/CT scanner, followed by a total-body PET/CT scan with the uEXPLORER scanner
  Arms: mCT/uEXPLORER

SUMMARY:
To determine the minimum scan duration for fluorine-18 positron-emitting radioactive isotope-fluorodeoxyglucose (18F-FDG) positron emission tomography (PET)/computed tomography (CT) scans performed on a total-body PET/CT scanner that results in non-inferior image quality to 18F-FDG PET/CT scans performed on a conventional PET/CT scanner. The subject population will be patients being staged for lung cancer, lymphoma, or melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign an informed consent form.
2. Ability to adhere to the study visit schedule and all protocol requirements.
3. Men and women ≥18 years of age.
4. Diagnosis or suspected diagnosis of lung cancer, melanoma or lymphoma.
5. Patients who have been referred for a PET/CT scan.

Exclusion Criteria:

1. Pregnant women.
2. Claustrophobia.
3. Any significant medical condition that in the opinion of the investigator would prevent the subject from participating and/or adhering to study related procedures or interfere with subject safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Minimum scan duration on a total-body PET/CT scanner for quality | One imaging visit up to two hours
  To determine the minimum scan duration for 18F-FDG PET/CT scans performed on a total-body PET/CT scanner that results in non-inferior image quality to 18F-FDG PET/CT scans performed on a conventional PET/CT scanner over 20 minutes.

SECONDARY OUTCOMES:
Minimum scan duration on a total-body PET/CT scanner for tumor recognition | One imaging visit up to two hours
  To determine the minimum scan duration for 18F-FDG PET/CT scans performed on a total-body PET/CT scanner that results in non-inferior tumor conspicuity to 18F-FDG PET/CT scans performed on a conventional PET/CT scanner over 20 minutes (with an additional 2 minutes of data used for optimization purposes).

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Nardo, MD, Principal Investigator — UC Davis Department of Radiology
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No